CLINICAL TRIAL: NCT04050670
Title: Effect of Injection Site on the Relative Bioavailability of a Single Dose of Tirzepatide in Subjects With Low and High Body Mass Indices
Brief Title: A Study of Tirzepatide at Different Injection Sites in Participants With Different Body Sizes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 17224; I8F-MC-GPHI (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-08-07; First posted 2019-08-08 (Actual); Results first posted 2023-03-24 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Healthy
MeSH Terms: interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tirzepatide - Upper Arm (Experimental): Participants received 5mg Tirzepatide by subcutaneous injection on upper arm.
  Interventions: Drug: Tirzepatide
- Tirzepatide - Thigh (Experimental): Participants received 5mg Tirzepatide by subcutaneous injection on thigh.
  Interventions: Drug: Tirzepatide
- Tirzepatide - Abdomen (Active Comparator): Participants received 5mg Tirzepatide by subcutaneous injection on abdomen.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Tirzepatide administered SC
  Other Names: LY3298176

SUMMARY:
The purpose of this study is to compare the amount of tirzepatide that gets into the blood stream and how long it takes the body to get rid of it, when injected under the skin of the upper arm and thigh compared to the abdomen. The study will be conducted in healthy males and females with different body sizes. The tolerability of tirzepatide will be evaluated and information about any side effects experienced will be collected. For each participant, the study will last about 20 weeks, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females of nonchildbearing potential as determined by medical history, physical examination, and other screening procedures
* Are between the body mass index (BMI) of 18.5 and 45.0 kilograms per meter squared (kg/m²), inclusive, at screening
* Are agreeable to receiving study treatment by injections under the skin

Exclusion Criteria:

* Have known allergies to tirzepatide or related compounds
* Have a personal or family history of medullary thyroid carcinoma or have multiple endocrine neoplasia syndrome type 2
* Have a history or presence of pancreatitis (history of chronic pancreatitis or idiopathic acute pancreatitis), elevation in serum amylase or lipase or gastrointestinal (GI) disorder (eg, relevant esophageal reflux or gall bladder disease) or any GI disease which impacts gastric emptying (eg, gastric bypass surgery, pyloric stenosis, with the exception of appendectomy) or could be aggravated by glucagon-like peptide-1 (GLP-1) analogs or dipeptidyl peptidase IV (DPP-IV) inhibitors
* Have a prior history of malignant disease(s) in the past 5 years prior to screening
* Smoke more than the equivalent of 10 cigarettes per day
* Is a known user of drugs of abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Inc, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was a washout period of at least 35 days between Tirzepatide injections.
Groups:
- Sequence 1: Participants received single dose of 5 milligram (mg) Tirzepatide by subcutaneous injection on upper arm in period 1, on thigh in period 2 and on abdomen in period 3.
- Sequence 2: Participants received single dose of 5 milligram (mg) Tirzepatide by subcutaneous injection on abdomen in period 1, on upper arm in period 2 and on thigh in period 3.
- Sequence 3: Participants received single dose of 5 milligram (mg) Tirzepatide by subcutaneous injection on thigh in period 1, on abdomen in period 2 and on upper arm in period 3.
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Started | 18 | 18 | 18
Received at Least One Dose of Study Drug | 18 | 18 | 18
Completed | 18 | 18 | 18
Not Completed | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Started | 18 | 18 | 18
Received at Least One Dose | 18 | 18 | 18
Completed | 18 | 18 | 18
Not Completed | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Started | 18 | 18 | 18
Received at Least One Dose | 18 | 17 | 18
Completed | 18 | 17 | 18
Not Completed | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- All Participants: Participants received 5mg Tirzepatide by subcutaneous injection administered through either upper arms or abdomen or thigh as per the dosing sequence.
Arm/Group | All Participants
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 54

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve of Tirzepatide From Time Zero to Infinity (AUC[0-∞])
Description: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve of Tirzepatide From Time Zero to Infinity (AUC[0-∞]) was evaluated.
Time Frame: Predose, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 336, 480 hours post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour * nanogram per milliliter (h*ng/mL)
Arm/Group | Tirzepatide - Abdomen | Tirzepatide - Upper Arm | Tirzepatide - Thigh
Number analyzed (Participants) | 54 | 54 | 53
Hour * nanogram per milliliter (h*ng/mL) | 112000 (24) | 111000 (21) | 106000 (22)
Statistical Analysis 1: Comparison: Tirzepatide - Abdomen vs Tirzepatide - Thigh; Test type: Non-Inferiority — A priori estimates for the 90% CI geometric least square means ratios of AUC(0-∞) for the thigh versus abdomen injection sites were from 0.80 to 1.25; Linear mixed effects model; Ratio of geometric least squares mean = 0.953, 90% CI 2-sided [0.935 to 0.970]
Statistical Analysis 2: Comparison: Tirzepatide - Abdomen vs Tirzepatide - Upper Arm; Test type: Non-Inferiority — A priori estimates for the 90% CI geometric least square means ratios of AUC(0-∞) for the upper arm versus abdomen injection sites were from 0.80 to 1.25; Linear mixed effects model; Ratio of geometric least squares mean = 0.990, 90% CI 2-sided [0.972 to 1.01]

2. Primary Outcome: PK: Maximum Concentration (Cmax) of Tirzepatide
Description: PK: Maximum Concentration (Cmax) of Tirzepatide was evaluated.
Time Frame: Predose, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 336, 480 hours post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per Millilitre (ng/mL)
Arm/Group | Tirzepatide - Abdomen | Tirzepatide - Upper Arm | Tirzepatide - Thigh
Number analyzed (Participants) | 54 | 54 | 53
Nanogram per Millilitre (ng/mL) | 603 (25) | 556 (23) | 520 (21)
Statistical Analysis 1: Comparison: Tirzepatide - Abdomen vs Tirzepatide - Thigh; Test type: Non-Inferiority — A priori estimates for the 90% CI geometric least square means ratios of Cmax for thigh versus abdomen injection sites were from 0.80 to 1.25; Linear mixed effects model; Ratio of geometric least squares mean = 0.862, 90% CI 2-sided [0.818 to 0.909]
Statistical Analysis 2: Comparison: Tirzepatide - Abdomen vs Tirzepatide - Upper Arm; Test type: Non-Inferiority — A priori estimates for the 90% CI geometric least square means ratios of Cmax for the upper arm versus abdomen injection sites were from 0.80 to 1.25; Linear mixed effects model; Ratio of geometric least squares mean = 0.921, 95% CI 2-sided [0.874 to 0.971]

ADVERSE EVENTS:
Time Frame: Up to 36 days
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Tirzepatide - Abdomen | Tirzepatide - Upper Arm | Tirzepatide - Thigh
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/54 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/54 | 0/53
Other Adverse Events (participants affected / at risk) | 37/54 | 31/54 | 23/53
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tirzepatide - Abdomen (N=54) | Tirzepatide - Upper Arm (N=54) | Tirzepatide - Thigh (N=53)
Abdominal distension (Gastrointestinal disorders) | 8 (8) | 10 (10) | 8 (8)
Constipation (Gastrointestinal disorders) | 4 (4) | 2 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 10 (11) | 11 (13) | 6 (7)
Eructation (Gastrointestinal disorders) | 3 (3) | 4 (5) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 20 (21) | 12 (12) | 11 (12)
Vomiting (Gastrointestinal disorders) | 9 (10) | 10 (10) | 4 (4)
Early satiety (General disorders) | 2 (2) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 13 (13) | 7 (7) | 3 (3)
Headache (Nervous system disorders) | 12 (14) | 8 (8) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-06-27): https://cdn.clinicaltrials.gov/large-docs/70/NCT04050670/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT04050670/SAP_001.pdf